CLINICAL TRIAL: NCT07032064
Title: Electrical and Hemodynamic Assessment of Pacing Modalities in Patients With Indications for Cardiac Resynchronization Therapy
Brief Title: Evaluation of Electrical and Hemodynamic Effects of Different Pacing Strategies in CRT Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Yixiu Liang, Professor, Chief Physician, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPP-Electro-Hemo
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure; CRT and/or ICD
Keywords: Cardiac resynchronization therapy;; Cardiac physiologic pacing；; Heart failure; Left bundle branch area pacing; Electrical resynchronization; Hemodynamic assessment
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of five pacing strategies in a Single-Arm CRT candidate cohort (Experimental): All enrolled patients will undergo sequential pacing at five ventricular sites during a single procedure: His bundle pacing (HBP), deep septal pacing (DSP), left ventricular septal pacing (LVSP), non-selective left bundle branch pacing (NS-LBBP), and selective left bundle branch pacing (SLBBP). Each pacing mode will be tested under identical physiological conditions in the same individual, and electrical and hemodynamic parameters will be recorded for comparative analysis. The order of pacing may be randomized or standardized according to protocol.
  Interventions: Procedure: Sequential ventricular pacing at five sites

INTERVENTIONS:
Procedure: Sequential ventricular pacing at five sites — This intervention involves sequential temporary pacing at five distinct ventricular sites within the same patient during a single electrophysiological study. The pacing sites include:His bundle pacing (HBP),Deep septal pacing (DSP),Left ventricular septal pacing (LVSP),Non-selective left bundle branch pacing (NS-LBBP),Selective left bundle branch pacing (SLBBP).
  Each pacing modality is tested under identical hemodynamic and electrophysiological conditions using a fixed output and AV delay. Electrical parameters and acute hemodynamic responses are recorded for each site. The study uses a within-subject crossover design, allowing direct intra-individual comparison of different pacing strategies in patients meeting standard CRT indications. No long-term device implantation is involved during this phase of the study.

SUMMARY:
Heart failure patients with delayed electrical activation of the heart often benefit from cardiac resynchronization therapy (CRT). However, traditional CRT using biventricular pacing is not effective in all patients. This study aims to evaluate the acute effects of pacing at different sites within the heart's conduction system-including His bundle pacing, deep septal pacing, left ventricular septal pacing, non-selective left bundle branch pacing, and selective left bundle branch pacing.

We will assess how these pacing strategies improve electrical synchrony and heart function by analyzing ECG parameters, such as QRS duration and QRS area, and measuring hemodynamic response using left ventricular pressure changes. The goal is to identify which pacing site provides the best improvement in heart performance. The study includes patients with left bundle branch block or intraventricular conduction delay, reduced heart function (ejection fraction <35%), and prolonged QRS duration (>150 ms).

This research may help improve the effectiveness of pacing therapy in heart failure patients who are not responding well to current CRT methods.

DETAILED DESCRIPTION:
This is a prospective, single-center, crossover study designed to evaluate the acute hemodynamic and electrical effects of pacing at five distinct sites within the conduction system in patients with heart failure and wide QRS complexes. Each participant will undergo temporary pacing at the His bundle, deep septal, left ventricular septal, non-selective left bundle branch, and selective left bundle branch sites.

Pacing sites will be confirmed by fluoroscopic guidance and intracardiac electrogram criteria, including stimulus-to-R' interval and QRS morphology. Hemodynamic response during each pacing mode will be assessed non-invasively using a Finometer device, which continuously measures beat-to-beat blood pressure and provides derived parameters of cardiac function.

The primary objective is to compare the relative hemodynamic benefits and electrical synchrony achieved at each pacing location, with the aim of optimizing lead placement strategies for conduction system pacing in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

NYHA class I to ambulatory IV despite optimized medical therapy for ≥3 months, LVEF ≤35%, and sinus rhythm with LBBB. LBBB was defined as QRS duration ≥130 ms, QS or rS in lead V1, broad/notched R waves in leads I, aVL, V5-V6, and absence of q waves in V5-V6

Exclusion Criteria:

second- or third-degree AV block, frequent PVCs, moderate-to-severe aortic stenosis, LV thrombus, or significant peripheral vascular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
QRSd | within 30 minutes per patient
  QRSd was measured from the onset to the end of the QRS complex
QRSa | within 30 minutes per patient
  QRSa was computed as the sum of the QRS area across three orthogonal vectorcardiographic leads reconstructed using the Kors transformation matrices
Hemodynamic Evaluation | within 30 minutes per patient
  Continuous non-invasive blood pressure was monitored using a Finometer device

CONTACTS AND LOCATIONS:
Overall Officials: Yixiu Liang, M.D., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: IPD could be requested by contacting the corresponding author via email after publication.